CLINICAL TRIAL: NCT03969628
Title: CARies DEtection in Children-Pelotas (CARDEC-PEL): Comparison of Two Methods of Caries Risk Assessment in Children
Brief Title: CARDEC-PEL: Comparison of Two Methods of Caries Risk Assessment in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Principal Investigator, Federal University of Pelotas
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PPGO 0030
Record Dates: First submitted 2019-05-29; First posted 2019-05-31 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Caries,Dental
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multivariate risk assessment group (ICCMS®) (Experimental): Multivariate risk assessment group (ICCMS®): multivariate caries risk assessment based on International Caries Classification and Management System (ICCMS™) guide
  Interventions: Diagnostic Test: ICCMS
- Simplified risk assessment group (dental caries experience) (Experimental): Simplified risk assessment group (dental caries experience): simplified caries risk assessment based on dental caries experience (WHO criteria)
  Interventions: Diagnostic Test: ICCMS

INTERVENTIONS:
Diagnostic Test: ICCMS — Risk caries assessment will consider ICCMS criteria

SUMMARY:
The aim of the study was to compare dental caries treatment and follow-up based on an elaborate and individualized assessment of caries risk in children, to a simpler risk assessment strategy by means of a double-blind randomized clinical trial of two years monitoring. Participants will be children from 7 to 11 years old, who pass through the screening of the Children's Clinic of the Faculty of Dentistry of the Federal University of Pelotas and fulfill the inclusion criteria. A randomized, stratified sample of approximately 250 children will be included in the study, one group will be composed of children undergoing dental caries-related treatment and maintenance, guided by an individualized and multivariate risk assessment, and another group of children treated based on dental caries experience alone in the deciduous and / or permanent dentition. Recruitment will begin at the beginning of 2019, and participants will be followed up for 24 months. Parents will respond to an anamnesis, 24-hour dietary recall, food frequency questionnaire, and oral and general health-related quality of life questionnaire, children will undergo a clinical examination to assess caries, according to the International Caries Detection and Assessment System (ICDAS) in its simplified form and evaluation of caries activity. Dental treatments and return intervals will be designated according to the individual risk of the patient detected in the initial approach according to the group. The study evaluations consist of baseline, 12 months and 24 months, data will be transferred to spreadsheets after the different phases of the study. Primary outcomes (number of dental surfaces requiring operative intervention) and secondary outcomes will be analyzed by Student's t test, quality of life and quality of life related to oral health, will be assessed at the beginning of the study and at the end of treatment, and compared between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 7 years months to 11 years;
* Children seeking dental treatment at the Pediatric dentistry university clinic in Pelotas (UFPel)

Exclusion Criteria:

* Medical and/or behavioral conditions that requires special considerations regarding management/treatment of the child

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 250 (Estimated)
Dates: Start 2019-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
New caries lesions | from baseline (first measurement) to 24months
  Incremental number of dental surfaces with operative treatment needs. This outcome will be assessed by the new caries lesions and / or progression of lesions previously diagnosed / treated and number of treated surfaces which will need restoration replacement, endodontic treatment or extraction after the treatment plan.

SECONDARY OUTCOMES:
Quality of life score | from baseline (first measurement) to 24months
  Impact on oral health related quality of life measured by a validated questionnaire (CPQ)

CONTACTS AND LOCATIONS:
Locations (1):
- Graduate Program in Dentistry, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menegaz AM, Oliveira TTDV, Braga MM, Raggio DP, Cenci MS, Mendes FM, Azevedo MS. Randomized clinical trial to evaluate two methods of caries risk assessment in schoolchildren: the CARDEC-PEL 04 study protocol. BMC Oral Health. 2021 Dec 18;21(1):654. doi: 10.1186/s12903-021-02010-3. PMID 34922527